CLINICAL TRIAL: NCT05046106
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Response Efficacy and Safety Study of MLC1501 in Patients With Stroke
Brief Title: MLC1501 Study Assessing Efficacy in STROke Recovery
Acronym: MAEStro
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Moleac Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFSA2019_01
Record Dates: First submitted 2021-09-02; First posted 2021-09-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Stroke, Ischemic; Strokes Thrombotic; Stroke Sequelae; Stroke, Cardiovascular; Stroke, Embolic; Stroke, Cryptogenic
Keywords: stroke; MLC1501; MAEStro; stroke recovery; neurorestoration
MeSH Terms: conditions — Stroke; Ischemic Stroke; Thrombotic Stroke; Myocardial Infarction; Embolic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 500-mg placebo capsule, 4 capsules twice a day for 24 weeks.
  Interventions: Other: Placebo
- MLC1501 Low-dose (Active Comparator): MLC1501 low-dose 500-mg capsule, 4 capsules twice a day for 24 weeks.
  Interventions: Drug: MLC1501
- MLC1501 High-dose (Active Comparator): MLC1501 high-dose 500-mg capsule, 4 capsules twice a day for 24 weeks.
  Interventions: Drug: MLC1501

INTERVENTIONS:
Drug: MLC1501 — Powdered extract of Radix astragali, Rhizoma chuanxiong, Radix angelica sinensis, Radix polygala
  Arms: MLC1501 High-dose; MLC1501 Low-dose
Other: Placebo — Caramel, chocolate brown, flavor (E_1982648), dextrin
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, dose-response study of MLC1501 in patients with stroke. Eligible participants will be randomized in a 1:1:1 ratio to orally receive MLC1501 low-dose twice a day, MLC1501 high-dose twice a day, or matching placebo for 24 weeks.

DETAILED DESCRIPTION:
A total of 540 patients will be included with approximately 180 participants randomized to each treatment arm. Randomization will be performed centrally and stratified according to the following factors at the time of randomization: NIHSS (8 to 12, 13 to 18), age (<65 years, ≥65 years) and received either intravenous or endovascular thrombolysis/thrombectomy (no, yes).

Efficacy clinical assessments will include mRS, FMA, ARAT, 10MWT, NIHSS, Barthel Index, EQ-5D-5L, MoCA, PROMIS-10, and occurrence of recurrent vascular event.

Each participant will undergo standard safety assessments including physical exam and laboratory parameters, and be observed for adverse events for the duration of the study. Electrocardiogram (ECG), hematology, clinical chemistry, coagulation, and urinalysis will be performed at specified intervals. The C-SSRS will be used to screen for suicidal ideation and behavior. Blood samples will be collected and stored for future studies on circulating compounds and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* 18 years old or older.
* Diagnosed with acute ischemic stroke with compatible brain imaging findings between 2 days to 7 days prior to inclusion. Patients who undergo intravenous or endovascular thrombolysis or thrombectomy must be considered stable for at least 24 hours post-procedure prior to inclusion.
* NIHSS total score of 8 to 18 (inclusive) at the time of inclusion with a combined score of at least 2 on the NIHSS motor items 5A or 5B and/or 6A or 6B.
* A candidate for active rehabilitation in the opinion of the treating physician.
* Able to comply with the requirements of the protocol and provide written informed consent by patient or legal representative before any study-specific procedure is performed.

Exclusion Criteria:

* Pre-stroke modified Rankin score of >1.
* Contraindication to any of the study procedures.
* Participation in another investigational drug or device trial within the past 30 days.
* Intake of warfarin in the past one week or expected to be on warfarin while in the study.
* Women who are pregnant, breastfeeding, of child-bearing potential or planning to become pregnant during the study. Menopausal/post-menopausal women without menstruation for 12 consecutive months or surgically sterilized women may be included. Intake of oral contraceptive pills or hormone replacement therapy is not allowed. Use of mechanical barriers, e.g., condom, intrauterine device, are allowed. Local contraception requirements for clinical trials should be followed.
* Any known food allergy or hypersensitivity to Astragalus membranaceus, Ligusticum chuanxiong, Polygala tenuifolia, Angelica sinensis, or members of the Fabaceae/Leguminosae family (e.g., legume, pea, bean), Polygalaceae family (e.g., milkwort, snakeroot), Apiaceae/Umbelliferae family (e.g., anise, caraway, carrot, celery, dill, parsley, parsnip), or Quillaja bark (soapbark).
* Evidence of other significant non-ischemic brain lesion which could affect long-term function or disability.
* Evidence of advanced medical condition that would affect study assessment and follow-up, such as cancer, renal failure, liver cirrhosis, severe dementia, or psychosis.
* Any other medical or psychiatric or cognitive condition which, in the study investigator's opinion, may jeopardize the patient by his/her participation in this study, may hamper his/her ability to complete procedures required in the study, affect study assessment and follow-up, or affect the validity of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 24 weeks
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 (no symptoms at all) to 5 (severe disability). A separate category of 6 is usually added for patients who expire.

SECONDARY OUTCOMES:
Fugl-Meyer motor Assessment (FMA) | 12, 24 weeks
Action Research Arm Test (ARAT) | 12, 24 weeks
Timed 10-Meter Walk Test (10MWT) | 12, 24 weeks
National Institute of Health Stroke Scale total and motor scores | 12, 24 weeks
  The maximum possible score is 42 (severe), with the minimum score being a 0 (no symptoms)
Barthel Index | 4, 12, 24, 36 weeks
EuroQol 5 Dimensions 5 Levels | 4, 12, 24, 36 weeks
  EQ5D-5L has 5 response levels: level 1 (no problems), 2 (slight), 3 (moderate), 4 (severe). Sometimes it is more convenient to dichotomies the levels into 'no problem's (level 1) and 'any problems' (level 2 to 5). In total, there are 3,125 possible unique health states defined by the EQ-5D-5L, with 11111 and 55555 representing the best and worst health states
Montreal Cognitive Assessment (MoCA) | 12, 24 weeks
Occurrence of recurrent vascular event | 24, 36 weeks
Patient Reported Outcome Measurement Information System - Global Health | 12, 24 weeks
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Columbia-Suicide Severity Rating Scale screen | 4, 12, 24, 36 weeks
  There are no specified clinical cutoffs for the C-SSRS due to the binary nature of the responses to items. When an item is endorsed, the clinician must pose follow-up inquiries to obtain additional information. The following can inform safety monitoring and treatment planning when patients endorse suicidal ideation, suicidal behavior, or both:
  * Suicidal ideation (Item endorsement: Yes; C-SSRS Categories 1-5)
  * Suicidal behavior (Item endorsement: Yes; C-SSRS Categories 6-10)
  * Suicidal ideation & behavior (Item endorsement: Yes; C-SSRS Categories 1-10)
Adverse events | up to 36 weeks
  Listing and calculating the number and percentage of subjects experiencing non-serious and serious adverse events for each dose cohort
modified Rankin Scale | 4, 12 and 36 weeks
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 (no symptoms at all) to 5 (severe disability). A separate category of 6 is usually added for patients who expire.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chen, BMBCh, MRCP, FAMS, FRCPE, Principal Investigator — Departments of Pharmacology and Psychological Medicine, National University of Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Once decided, only anonymized IPD may be shared with other collaborative stroke trials consortiums.